CLINICAL TRIAL: NCT01463787
Title: Comparison of Outcomes of Two Approaches in Microsurgical Varicocelectomy in Chinese Infertile Males: A Prospective Randomized, Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Feng Pan (Other)
Responsible Party: Sponsor-Investigator, Feng Pan, Clinical Attending Doctor, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FPan
Record Dates: First submitted 2011-10-26; First posted 2011-11-02 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Varicocele
Keywords: Infertility; varicocelectomy; microsurgery; Chinese men; pregnancy rate
MeSH Terms: conditions — Varicocele; Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inguinal group (Experimental)
  Interventions: Procedure: microsurgical varicocelectomy in inguinal approach
- sub-inguinal group (Active Comparator)
  Interventions: Procedure: microsurgical varicocelectomy in subinguinal approach

INTERVENTIONS:
Procedure: microsurgical varicocelectomy in inguinal approach — In inguinal approach, the incision, which was about 3cm, was made two fingers up the pubic symphysis, from external inguinal rings parallel to the inguinal ligament.
  Arms: inguinal group
Procedure: microsurgical varicocelectomy in subinguinal approach — In subinguinal approach, the incision was about 3 cm horizontal and 1 cm below the external inguinal ring.
  Arms: sub-inguinal group

SUMMARY:
Varicocele is the most common surgical disease which could lead to male infertility. It is found in approximately 15% adult males, and in about 40% infertile males. And the incidence is up to 80% in secondary infertility. In the past, there was continuous controversy over whether a varicocele repair could improve fertility. But at present, researches are coming to a consensus on the indication of varicocelectomy. Several researches manifest that the microsurgery of varicocele could have the effect of the highest spontaneous pregnancy and lowest complications rate after surgery. Microsurgical varicocelectomy includes two approaches, inguinal and subinguinal. Each one has its advantages and disadvantages. There are few studies which make direct comparison between the two methods in microsurgical varicocelectomy, especially in China. Operators have made decisions on the basis of their own experience and skills. In this study, the investigators compare the postoperative spontaneous pregnancy and complications rates in two approaches in microsurgical varicocelectomy for Chinese infertile men in their hospital.

DETAILED DESCRIPTION:
Outcome Measures

Before surgery, all patients were diagnosed by physical examination and testified by color Doppler ultrasound. And one trained nurse documented the patients' age, left unilateral or bilateral and the grade of varicocele, and the grade of the more serious side was noted when handled with bilateral ones. During surgery, the duration of surgery was documented. After surgery, a Visual Analogue Scale (VAS) was used to assess the introperative pain after anesthesia recovery and the amount of postoperative pain one month postoperatively by another trained nurse. And the patients whose pain scores > 3 and/or who claimed pain were prescribed with ibuprofen sustained-release capsules (China SmithKline Pharmaceutical Company, Tianjing, China) (0.3g) (ISRC) every 12h on the surgical day (since 2h postoperatively) and only if necessary on the following days (no patient claimed that he had gastrointestinal ulcer history or allergic history of relative drug). Parents were told to write down on a provided form how many times they gave medicine postoperatively. Patients were followed with visits 1 month, 3, 6 and 12 months after surgery, and were encouraged to visit the clinic anytime when they had any complaint in this period. The semen analyses were conducted in the 3, 6 and 12 months in the follow-up. The recurrence or hydrocele formation was testified by color Doppler ultrasound (with/without detected by physical examination) by the same doctor who did the preoperative examination. And this doctor and two nurses mentioned above were all unaware of the patients' groups.

ELIGIBILITY:
Inclusion Criteria:

1. Primary infertility (more than 1 year)
2. Serum hormone was normal (FSH, LH, T and PRL)
3. Semen analysis which was taken within 3-7 days of abstinence was abnormal for at least twice, and at least 1 month apart (the value of sperm density was less than 20 million per ml, and/or sperm motility a+b was less than 50%, according to the 4th WHO criteria)
4. All varicocele was diagnosed by physical examination and testified by color Doppler ultrasound
5. Patients' spouse was healthy in reproduction or had some curable generational diseases

Exclusion Criteria:

1. Secondary infertility
2. Men with subclinical varicocele or normal semen analyses
3. Having some other surgical diseases, such as genital tract infection or deformity
4. Having some congenital diseases, such as Klinefelter and Y chromosome deficiency
5. Having some endocrine diseases, such as Kallmann, abnormality in pituitary gland, hyperthyroidism, hypercorticoidism, and so on
6. Patients' spouse had some diseases that made them unable to carry out spontaneous pregnancy, such as tubal obstruction or ovulatory failure.

Ages: 20 Years to 46 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
pregnancy | within the 12-24 months postoperative period
  Postoperative spontaneous pregnancy is considered to be the best indicator to assess fertility status.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Maternity and Child Healthcare Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China